CLINICAL TRIAL: NCT07306000
Title: Effects of Close Collaboration With Parents Intervention on NICU Care Environments and Long-term Development of Preterm Infants: a Pilot Study
Brief Title: Pilot Study: Effects of CCP Intervention on NICU Environment and Preterm Infants Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Liisa Lehtonen, Professor, Turku University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PilotStudy/2025
Record Dates: First submitted 2025-11-26; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Preterm Infant Development; Preterm Infant Health
Keywords: close collaboration with parents; family-centered care

STUDY DESIGN:
Intervention Model Description: 1. Unidirectional crossover design within one center: self-controlled comparison (pre- vs. post-intervention)
  2. Stepped-wedged cluster study across multi-centers: parallel comparison (NICU A post-intervention vs. NICU B/C pre-intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): Prior to the implementation of the Close Collaboration with Parents (CCP) training program, staff provide routine care according to standard NICU practices.
- Post-intervention (Experimental): After the implementation of the CCP training program, all NICU staff participate in the intervention, applying the learned practices to include parents in the care of their infants in the NICU.
  Interventions: Behavioral: Close Collaboration with Parents training

INTERVENTIONS:
Behavioral: Close Collaboration with Parents training — The Close Collaboration with Parents is an educational intervention for neonatal health care staff. The "train the trainer" model is used in the implementation so that the training team trains local mentors in each NICU, who then mentor the other neonatal health care staff. Local mentors are chosen from the neonatal health care team (nurses, doctors, or psychologists) working in the NICU. The learning process of neonatal health care teams includes completing the e-learning module and bedside practices combined with reflection on the practice experience with a local mentor. The final goal is to improve the family-centered care culture of the NICU by developing the skills of the neonatal health care team to communicate and collaborate with parents and to provide support for parenting.
  Arms: Post-intervention

SUMMARY:
Close Collaboration with Parents intervention is an evidence-based educational intervention for the entire multi-professional staff of neonatal intensive care units (NICUs). The goal of the intervention is to strengthen partnership between staff and parents, enhance parental participation in infant care. There are no studies yet about the effects of the Close Collaboration with Parents intervention on the long-term neurodevelopment and socio-emotional development of very preterm infants and their interaction with their parents. Accordingly, a multicenter cluster randomized controlled trial is planned. Prior to initiating this large-scale study, it is essential to validate the measurement instruments. Therefore, a pilot study will be conducted to assess their feasibility and to determine the appropriate sample size.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born below 32 weeks of gestation and/or weighing < 1500 g who receive long-term follow-up at each study site.

Exclusion Criteria:

* the infant has any major anomalies
* the infants are triplets or higher order
* the infant's condition is critical and the survival is uncertain
* the parents cannot understand the informed consent form in Korean or in Japanese

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Auditory environment: parent and adult speech | Once a week, for 24 hours (every 7 days, up to 40 weeks of postmenstrual age)
  The quantity of adult speech is recorded and analyzed. The quantity of adult speech includes the duration (minutes per hour), number of words (per hour), syllables (per hour), and phonemes (per hour). The recording is done with a commercial recording device. The microphone is placed in the incubator or infant cot. The data analyses are performed using ALICE, an open-source tool to count words, syllables, and phonemes.
Auditory environment: sound level and its variation | Once a week, for 24 hours (every 7 days, up to 40 weeks of postmenstrual age)
  The sound level includes sound pressure (dB) and its variation. The main focus of this measurement is to detect a sudden change in the sound pressure caused by alarms and other activities which are a common source of stress in a NICU environment. The recording is done with a sound level detector, a different device from that for speech recording. The microphone is placed in the incubator or infant cot. The data analyses are performed using a one-minute resolution of the recording regarding the average, maximum and minimum and 5 and 95 percentiles of the sound level.
Sensitive care: sleep quality and quantity | Once a week, for 24 hours (every 7 days, up to 40 weeks of postmenstrual age)
  The artificial intelligence-based algorithm tool to analyze infant behavior with a camera captured image will be used to classify infant state into six categories: Non-REM (rapid eye movement) sleep, REM (rapid eye movement) sleep, drowsy, quiet awake, active awake, and crying. In addition, caretaking and procedures will be recorded and scored. The diary data is used to get information of the times the infants is not under the camera image like during skin-to-skin contact. The camera is custom-designed with the connection to a local computer. The night-vision camera works well also in a dimmed light environment. The module can be used for both infants in an incubator and in an open bed.
Parents' presence and parent-infant skin-to-skin contact | Once a week, for 24 hours (every 7 days, up to 40 weeks of postmenstrual age)
  Parents' presence is defined as their presence beside their infant or at least in the same room with the infant. Parent-infant skin-to-skin contact is defined as the infant being held by the parent on the bare chest, with only a diaper and a cap if necessary.
  The duration of parents' presence and parent-infant skin-to-skin contact will be recorded using a modified Parent-Infant Closeness Diary. Parents or staff indicate the specific items by drawing a line. The caretaking includes hands-on care and holding, breastfeeding and bottle feeding of the infant. The start and the end times should be put in 5-minute increments.
Type of enteral feeding | Once a week, for 24 hours (every 7 days, up to 40 weeks of postmenstrual age)
  The amount of enteral feeding divided into 4 categories, fresh breast milk, refrigerated/frozen breast milk, donated breast milk, and formula milk will be collected per day. Both the absolute amount of milk and its proportion of the total enteral nutrition will be calculated. We hypothesize that the infants will receive more fresh maternal milk after the intervention.
Body weight | every 7 days, from enrollment to the NICU discharge (up to 40 weeks of postmenstrual age), 1 month of corrected age, 6 months of corrected age, 18 months of corrected age, and 36 months
  The body weight of the participated infant, and its percentile/Z-score based on the standardized growth curve (Fenton 2025 and National growth curve) will be collected.

SECONDARY OUTCOMES:
Breastfeeding | between 36+0 and 36+6 weeks of postmenstrual age (7 days), and between 7 and 1 day before the day of NICU discharge (7 days)
  The frequency (times per day) and proportion (% of total feeding number per day) of breastfeeding will be recorded between 36+0 and 36+6 weeks of postmenstrual age and between 7 and 1 day before the day of NICU discharge. Then the average frequency and proportion of breastfeeding at 36 weeks of postmenstrual age and at NICU discharge will be calculated.
Parents' parenting self-efficacy | at 36 weeks of postmenstrual age, at the day of NICU discharge (up to 40 weeks of postmenstrual age), and 1 month of corrected age
  The questionnaire consists of 26 questions about the parenting self-efficacy. Each question is rated by parents using a Likert scale from 1 (fully disagree) to 6 (fully agree).
Length of stay and PMA at discharge | at the day of NICU discharge (up to 40 weeks of postmenstrual age)
  The hospitalization duration and the postmenstrual age (PMA) at NICU discharge will be collected from the medical records.
Brain MRI | at the term age, between 37+0 and 41+6 weeks of postmenstrual age
  The brain MRI will be taken at the term age, between 37+0 and 41+6 weeks of postmenstrual age or shortly before the NICU discharge. The brain MRI image will be evaluated using a standardized scoring system, that consists of six items for white matter injury and seven for gray matter injury. The total score is 17 for white matter and 22 for gray matter and cerebellum. A higher score indicates better brain development. The severity of the injury is defined using the total score for white and gray matter, respectively.
Parent-infant interaction: eye movement and behavior tracking | at 6 months of corrected age, for 10 minutes
  The measurements will be done during a structured test situation. The mother or father and the child are positioned face-to-face at a table and engaged with a standardized set of toys for 10 minutes. The parent will wear glasses with an eye tracker and a camera. The child will not wear such devices due to the high rates of data attrition for child-held devices. Infant face-looking will be analyzed using a deep neural network based on the video data recorded by the parent's glasses. Parent's face-looking behavior will also be extracted from the eye tracking and video data recorded by the parent's glasses. Parent reactions to child face-looking (facial and vocal) will be obtained from a separate video and audio recording, using automatic tools.
Cry diary | at 6 months of corrected age, for 3 days
  The duration of the infants crying at home will be recorded using the Cry Diary. The parents record baby's state to 6 categories (sleeping, awake & happy, awake & fussy, awake & crying, feeding, not sure) and parents' action to 3 categories (holding the baby, transport, baby care) with 5-minute accuracy using the Cry Diary for 3 consecutive days, shortly before the 6 months corrected age follow-up visit.
Infant Behavior Questionnaire-Revised (IBQ-R) | at 6 months of corrected age
  The IBQ-R has 191 items in which parents rate their infant's behavior over the past one to two weeks on a 7-point Likert scale (1 = never, 7 = always) based on the frequency of the observed behavior. If a behavior was not observed, parents mark it as "not applicable". The items form three broad temperament dimensions with subscales: Surgency/Extraversion (Approach, Vocal Reactivity, High Intensity Pleasure, Smiling and Laughter, Activity Level), Negative Affectivity (Perceptual Sensitivity, Sadness, Distress to Limitations, Fear, Falling Reactivity), Orienting/Regulatory Capacity (Low Intensity Pleasure, Cuddliness, Duration of Orienting, Soothability). The IBQ-R has shown predictive validity for later child temperament and behavioral outcomes.
Early Childhood Behavior Questionnaire (ECBQ) | at 18 months of corrected age
  The ECBQ consists of 201 items and has the same 7-point scale as the IBQ-R. It measures three broad dimensions of temperament, each with multiple subscales: Surgency/Extraversion (Activity Level, High-Intensity Pleasure, Sociability, Impulsivity, Approach, Shyness), Negative Affectivity (Fear, Frustration, Discomfort, Sadness, Soothability), Effortful Control (Attention Focusing, Cuddliness, Inhibitory Control, Low-Intensity Pleasure, Perceptual Sensitivity. The ECBQ has shown predictive validity for children's later emotional and behavioral regulation.
Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) | at 18 months of corrected age and 3 years of age
  Bayley scale scores for each development areas (cognitive, language, motor) score range : 0-200 above average (1 to -2 standard deviation, score 116-130) average (1 to -1 standard deviation, score 85-115) below average (1 to -2 standard deviation, score 84-70) well below average (<-2 standard deviation, scores < 70).
Infant Toddler Social Emotional Assessment (ITSEA) | at 18 months of corrected age and 3 years of age
  The ITSEA is a screening method for infants between 12 and 36 months of age to predict their future social and emotional problems. It has 170 items, each rated from 0 (not true/rarely) to 2 (very true/often).

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (2):
  - Nagano Children's Hospital, Matsumoto, Nagano
  - Kyoto University Hospital, Kyoto
- Korea University Anam Hospital NICU, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
A decision has not yet been made regarding whether to share individual participant data or not. Because individual participant data contains a large amount of metric data and personal developmental outcomes, the researchers will discuss this matter further before making a decision.